CLINICAL TRIAL: NCT01243554
Title: Exercise Training in Pregnancy. Good for the Mother - Good for the Child?
Brief Title: Exercise Training in Pregnancy for Obese Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Norwegian School of Sport Sciences (Other); Karolinska Institutet (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ETiP-Ob
Record Dates: First submitted 2010-09-06; First posted 2010-11-18 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2018-06

CONDITIONS: Pregnancy; Obesity
Keywords: Exercise training; Pregnancy; Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): Supervised exercise training at the hospital during pregnancy: the women will attend at least 2 weekly sessions consisting of aerobic exercise (walking on treadmills), strength training (for upper body, back, abdomen and legs) as well as pelvic floor muscle exercises. Each session is 60 minutes and lead by a physiotherapist or experienced exercise physiologist. The women will also go through motivational interviewing sessions throughout the intervention period and are encouraged to do home exercise training in addition to the exercise at the hospital
  Interventions: Behavioral: Exercise
- Control (No Intervention): Usual care as provided by the health services in Norway. The investigators will not advice the women to be inactive

INTERVENTIONS:
Behavioral: Exercise — Exercise training at the hospital
  Other Names: Training
  Arms: Exercise training

SUMMARY:
Observational studies demonstrate that overweight in pregnancy is a risk factor for adverse pregnancy outcomes as fetal macrosomia, prolonged labor, low Apgar score, shoulder dystocia, nerve plexus injuries, increased proportion of instrumental deliveries and perineal ruptures. There is a 2.6 fold risk for gestational diabetes mellitus (fourfold in morbidly obese women) and a recent study has shown that fetuses of obese mothers develop insulin resistance in uterus.

Main aims of this study are to assess if regular exercise in pregnancy among obese women can prevent or influence weight gain; impaired cardiac function in mother and fetus/newborn; impaired vascular function in mother; insulin resistance/sensitivity; body composition in mother and offspring; lumbopelvic pain; urinary and/or fecal incontinence; prolonged labor

DETAILED DESCRIPTION:
Women with a self-reported pre-pregnancy BMI of 28 or more will be eligible for our study. Woman are eligible if they are 18 years or older, with a singleton live fetus at an early (week 12-14) ultrasound scan. Exclusion criteria are pregnancy complications with high risk for preterm labour or diseases that could interfere with participation.

Primary outcome measure is weight increase based on weight measured at 14 weeks and immediately before labour. Assessments are done at baseline at 14 (12-18) weeks of pregnancy, and again in week 38, as well as 3 months postpartum. Some measurements are also done at other points in time. The maternal secondary outcome measurements include fasting glucose, glucose tolerance assessed by 2-h, 75 mg per-oral glucose tolerance test, insulin resistance assessed by HOMA-IR, weight, height, body composition estimated by skinfold measurements in pregnancy and by dual energy x-ray absorptiometry postpartum, blood markers, lumbopelvic pain, urin- and fecal incontinence, quality of life, psychological wellbeing, depression, and diet.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pregnancy body mass index of 28 or more
* 18 years or more
* singleton live fetus at the routine ultrasound scan

Exclusion Criteria:

* high risk for preterm labor or diseases that could interfere with participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-09; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Weight gain during pregnancy | From 14 weeks pregnancy to delivery
  Measured in kg

SECONDARY OUTCOMES:
Fasting glucose | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  Blood samples to determine the fasting glucose after an overnight fast (>10 hours)
Glucose tolerance | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  2 hour 75 mg per-oral glucose tolerance test. Gestational diabetes is diagnosed as fasting glucose = or > 6.9 mmol/L or 2h concentration = or > 7.8 mmol/L.
Insulin resistance | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  Homeostasis model assessment (HOMA-IR)
Body composition | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  Skinfold measurements, done by an experienced investigator using Harpenden kaliper. At the 3 months postpartum testing, also dual energy x-ray absorptiometry (DEXA scan) will be used.
Blood markers for cardiovascular disease | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  Inflammation markers, cytokines (leptin, resistin, adiponectin, tnf-alfa). Blood will be collected and stored for later analyses.
Lumbopelvic pain | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  Clinical assessment (active straight leg raising, pelvic provocation test), and validated questionnaire.
Urin- and fecal incontinence | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  Pelvic floor muscle function will be assessed by clinical assessment and by 2D and 3D ultrasound. The prevalence and severity of urin- and fecal incontinence will also be assessed by a validated questionnaire
Quality of life | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  Validated questionnaire
Sleep | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  Epworth sleepiness scale
Physical activity | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  Level of physical activity will be assessed by activity registration (armbands) and by validated questionnaires
Diet | From 14 weeks pregnancy to 38 weeks pregnancy and also at 3 months postpartum
  Validated questionnaire: Norkost
Offspring birth weight, length and head circumference | At delivery
  As recorded by the hospital
Delivery complications | At delivery
  Vaginal or caesarean delivery, and recorded complications during the delivery
Markers of inflammation and metabolism in cord blood | At delivery
  Cord blood will be sampled and stored for later analysis of relevant markers of inflammation and metabolism (including resistin, leptin, adiponectin)

CONTACTS AND LOCATIONS:
Overall Officials: Trine T Moholdt, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Garnaes KK, Morkved S, Salvesen O, Moholdt T. Exercise Training and Weight Gain in Obese Pregnant Women: A Randomized Controlled Trial (ETIP Trial). PLoS Med. 2016 Jul 26;13(7):e1002079. doi: 10.1371/journal.pmed.1002079. eCollection 2016 Jul. PMID 27459375
- [Result] Garnaes KK, Nyrnes SA, Salvesen KA, Salvesen O, Morkved S, Moholdt T. Effect of supervised exercise training during pregnancy on neonatal and maternal outcomes among overweight and obese women. Secondary analyses of the ETIP trial: A randomised controlled trial. PLoS One. 2017 Mar 21;12(3):e0173937. doi: 10.1371/journal.pone.0173937. eCollection 2017. PMID 28323893
- [Result] Garnaes KK, Morkved S, Salvesen KA, Salvesen O, Moholdt T. Exercise training during pregnancy reduces circulating insulin levels in overweight/obese women postpartum: secondary analysis of a randomised controlled trial (the ETIP trial). BMC Pregnancy Childbirth. 2018 Jan 8;18(1):18. doi: 10.1186/s12884-017-1653-5. PMID 29310617
- [Result] Nyrnes SA, Garnaes KK, Salvesen O, Timilsina AS, Moholdt T, Ingul CB. Cardiac function in newborns of obese women and the effect of exercise during pregnancy. A randomized controlled trial. PLoS One. 2018 Jun 1;13(6):e0197334. doi: 10.1371/journal.pone.0197334. eCollection 2018. PMID 29856768
- [Result] Garnaes KK, Helvik AS, Stafne SN, Morkved S, Salvesen K, Salvesen O, Moholdt T. Effects of supervised exercise training during pregnancy on psychological well-being among overweight and obese women: secondary analyses of the ETIP-trial, a randomised controlled trial. BMJ Open. 2019 Nov 21;9(11):e028252. doi: 10.1136/bmjopen-2018-028252. PMID 31753866
- [Derived] Moholdt T, Garnaes KK, Vik IP, Morkved S, Salvesen KA, Ingul CB. Cardiovascular effects of exercise training in pregnant people with a high body mass index: secondary results from a randomised controlled trial (ETIP). BMJ Open Sport Exerc Med. 2024 Nov 21;10(4):e002099. doi: 10.1136/bmjsem-2024-002099. eCollection 2024. PMID 39610995
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Ingul CB, Loras L, Tegnander E, Eik-Nes SH, Brantberg A. Maternal obesity affects fetal myocardial function as early as in the first trimester. Ultrasound Obstet Gynecol. 2016 Apr;47(4):433-42. doi: 10.1002/uog.14841. Epub 2016 Mar 14. PMID 25761057
- [Derived] Moholdt TT, Salvesen K, Ingul CB, Vik T, Oken E, Morkved S. Exercise Training in Pregnancy for obese women (ETIP): study protocol for a randomised controlled trial. Trials. 2011 Jun 17;12:154. doi: 10.1186/1745-6215-12-154. PMID 21682869